CLINICAL TRIAL: NCT01388621
Title: PROVE A Randomized Phase II Trial of Standard Carboplatin-based Chemotherapy With or Without Panitumumab in Platinum-sensitive Recurrent Ovarian Cancer
Brief Title: Carboplatin-based Chemotherapy With or Without Panitumumab in Platinum-sensitive Recurrent Ovarian Cancer
Acronym: PROVE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: WiSP Wissenschaftlicher Service Pharma GmbH (Other)
Collaborators: ClinAssess GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMIHO-008/2009_AG56; 2010-018849-59 (EudraCT Number)
Record Dates: First submitted 2011-05-17; First posted 2011-07-06 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; fallopian cancer; recurrent; platinum-sensitive; KRAS-Wildtype
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — Panitumumab; liposomal doxorubicin; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental arm (A): (Experimental): Caelyx 30 mg/m² d1 Carboplatin AUC 5 d1 Panitumumab 6 mg/kg/KG d1 + 15 q4w until progressive disease or for a max. of 6 cycles
  OR
  Gemcitabine 1000 mg/m² d1 + 8 Carboplatin AUC 4 d1 Panitumumab 9 mg/kg/KG d1 q3w until progressive disease or for a max. of 6 cycles
  The backbone chemotherapy (Caelyx or Gemcitabine-based) is specified by the investigator before randomization of a patient.
  Interventions: Drug: Panitumumab; Drug: pegylated liposomal doxorubicin (PLD); Drug: Carboplatin; Drug: Gemcitabine
- Standard arm (B): (Active Comparator): Caelyx 30 mg/m² d1 Carboplatin AUC 5 d1 q4w until progressive disease or for a max. of 6 cycles
  OR
  Gemcitabine 1000 mg/m² d1 + 8 Carboplatin AUC 4 d1 q3w until progressive disease or for a max. of 6 cycles
  The backbone chemotherapy (Caelyx or Gemcitabine-based) is specified by the investigator before randomization of a patient.
  Interventions: Drug: pegylated liposomal doxorubicin (PLD); Drug: Carboplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Panitumumab — Panitumumab 6 mg/kg/BW d1 + 15 q4w until progressive disease or for a max. of 6 cycles In case of CR, PR or SD at the end of the combination treatment in experimental arm, panitumumab monotherapy is to be continued with 9 mg/kg/BW d1 q3w until time of tumor progression or up to a maximum of 6 months.
  Other Names: Vectibix
  Arms: Experimental arm (A):
Drug: pegylated liposomal doxorubicin (PLD) — pegylated liposomal doxorubicin (PLD) 30 mg/m² d1 q4w until progressive disease or for a max. of 6 cycles
  Other Names: Caelyx
Drug: Carboplatin — Carboplatin AUC 5 d1 q4w until progressive disease or for a max. of 6 cycles
  Other Names: multiple generics in existence
Drug: Gemcitabine — gemcitabine 1000 mg/m² d1 + 8 q3w until progressive disease or for a max. of 6 cycles
  Other Names: Gemzar
Drug: Carboplatin — Carboplatin AUC 4 d1 q3w until progressive disease or for a max. of 6 cycles
  Other Names: multiple generics in existence
Drug: Panitumumab — Panitumumab 9 mg/kg/BW d1 q3w until progressive disease or for a max. of 6 cycles In case of CR, PR or SD at the end of the combination treatment in experimental arm, panitumumab monotherapy is to be continued with 9 mg/kg/BW d1 q3w until time of tumor progression or up to a maximum of 6 months.
  Other Names: Vectibix
  Arms: Experimental arm (A):

SUMMARY:
The purpose of this trial is to estimate the therapeutic efficacy of the experimental targeted regimen including the EGFR antibody panitumumab (in combination with carboplatin and either pegylated liposomal doxorubicin or gemcitabine) in relation to the respective standard combination in patients with a KRAS wildtype with platinum-sensitive recurrent ovarian cancer. It is expected that the progression free survival rate at 12 months is improved by the targeted regimen.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with pretreated epithelial ovarian cancer, primary peritoneal carcinomatosis or fallopian tube cancer with histological confirmation of the tumor
* Wild-type k-ras status
* Patients must have pretreated platinum-sensitive ovarian cancer with recurrence more than 6 months after completion of a platinum-containing regimen
* Presence of at least one measurable or non-measurable disease (e.g. malignant ascites) following RECIST criteria by radiologic evaluation OR histological confirmation of recurrence by biopsy. The presence of non-measurable lesions only requires in addition a 2-fold increase of CA-125 elevation above normal lab value (confirmed by two measurements).
* No more than 2 prior treatment regimens for these epithelial cancers
* Age > 18 years.
* ECOG Performance Status of 0 or 1
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

  * Hemoglobin > 9.0 g/dl
  * Leukocyte count >3.000/mm3 ; absolute neutrophil count (ANC) >1.500/mm3
  * Platelet count ≥ 100.000/μl
  * Total bilirubin < 1,0 times the upper limit of normal
  * ALT and AST < 2,5 x upper limit of normal (< 5 x upper limit of normal for patients with liver involvement of their cancer)
  * Alkaline phosphatase < 4 x ULN
  * PT-INR/PTT < 1.5 x upper limit of normal [Patients who are being therapeutically anticoagulated with an agent such as coumarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists.]
  * Serum creatinine < 1.5 x upper limit of normal and creatinine clearance > 50 ml/min.
  * Magnesium ≥ lower limit of normal; calcium ≥ lower limit of normal
* Signed and dated informed consent before the start of specific protocol procedures.

Exclusion Criteria:

* Clinically significant cardiovascular disease (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before enrolment.
* History of interstitial lung disease, e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan.
* History of HIV infection or chronic hepatitis B or C
* Active clinically serious infections (> grade 2 NCI-CTC version 3.0)
* Pre-existing neuropathy > grade 1 (NCI CTCAE), except for loss of tendon reflex
* Prior radiological or clinical evidence of CNS metastases including previously treated, resected, or asymptomatic brain lesions or leptomeningeal involvement by head CT scan or MRI
* Patients with seizure disorder requiring medication (such as steroids or anti-epileptics)
* History of organ allograft
* Patients with evidence or history of bleeding diathesis
* Patients undergoing renal dialysis
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry.
* Patients in a closed institution according to an authority or court decision
* Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study

Excluded therapies and medications, previous and concomitant:

* Anticancer chemotherapy within 4 weeks prior to study entry.
* Prior anti-EGFR therapy
* Radiotherapy during study or within 4 weeks of start of study drug. (Palliative radiotherapy of non-target lesions will be allowed) and prior radiotherapy of > 25% of the bone marrow
* Major surgery within 4 weeks of start of study
* Autologous bone marrow transplant or stem cell rescue within 12 months of study
* Investigational drug therapy outside of this trial during or within 4 weeks of study entry
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate after 12 months. | 12 month
  PFS is defined as the time from randomisation to the time of disease progression or relapse (according to RECIST, not CA-125 only!) or death, or to the date of last tumor assessment without any such event (censored observation).

SECONDARY OUTCOMES:
Duration of Tumor-Response | Duration of Therapy (Therapy is planned for 6 cycles of 3 resp. 4 weeks each, shorter or longer durations are possible)
  according to RECIST, including measurable disease patients only, and including patients with CA-125 defined disease as well
Progression-free survival | End of Follow-up (up to 1 year)
Overall survival | End of Follow-up (up to 1 year)
Maximum toxicity resp. AE grade per patient per toxicity resp. AE during therapy | Duration of Therapy (Therapy is planned for 6 cycles of 3 resp. 4 weeks each, shorter or longer durations are possible)
  Toxicities resp. (S)AE during therapy will be documented, reported and analyzed according to NCI CTC 3.0 with special focus on skin toxicity.
  Results are given as maximum grade per patient per toxicity resp. AE during therapy.
Tumor Response Rate | Duration of Therapy (Therapy is planned for 6 cycles of 3 resp. 4 weeks each, shorter or longer durations are possible)
  according to RECIST, including measurable disease patients only, and including patients with CA-125 defined disease as well

CONTACTS AND LOCATIONS:
Overall Officials: Jalid Sehouli, MD (Prof. Dr. med.), Principal Investigator — Frauenklinik Charité - Universitätsmedizin Berlin Campus Virchow-Klinikum
Locations (18):
- Germany (18):
  - Praxis Dr. Oettle, Friedrichshafen, Baden-Wurttemberg
  - Stauferklinikum Schwäbisch Gmünd, Mutlangen, Baden-Wurttemberg
  - Carl-Thiem-Klinikum Cottbus Frauenklinik, Cottbus, Brandenburg
  - Praxis Dr. Heinrich, Fürstenwalde, Brandenburg
  - Tagesklinik Altonaer Strasse, Hamburg, Hamburg
  - MVM mbH Onkologische Schwerpunktpraxis Leer, Leer, Lower Saxony
  - Universitätsfrauenklinik am Klinikum Südstadt, Rostock, Mecklenburg-Vorpommern
  - Medizinisches Zentrum Bonn-Friedensplatz, Bonn, North Rhine-Westphalia
  - Klinikum Chemnitz Frauen- und Kinderklinik, Chemnitz, Saxony
  - Martin-Luther-Universität Halle-Wittenberg Zentrum für Frauenheilkunde und Geburtshilfe, Halle, Saxony-Anhalt
  - Klinikum Magdeburg, Magdeburg, Saxony-Anhalt
  - Praxisklinik Frauenheilkunde, Berlin, State of Berlin
  - Helios Klinikum Berlin - Buch, Berlin, State of Berlin
  - Frauenklinik Charité - Universitätsmedizin Berlin Campus Virchow-Klinikum, Berlin, State of Berlin
  - Ev. Waldkrankenhaus Spandau, Berlin, State of Berlin
  - Praxis Dr. Schilling / Till / Kohn FÄ f. Gynäkologie u. Geburtshilfe, Gynäkol.-Onkol. Schwerpunktpraxis, Berlin
  - Gynäkologische Praxis Dr. med. Ruhmland, Berlin
  - Park-Klinik Weißensee, Berlin